CLINICAL TRIAL: NCT04964934
Title: A Phase III, Double-blind, Randomised Study to Assess Switching to AZD9833 (a Next Generation, Oral SERD) + CDK4/6 Inhibitor vs Continuing Aromatase Inhibitor (Letrozole or Anastrozole)+ CDK4/6 Inhibitor in HR+/HER2-MBC Patients With Detectable ESR1Mutation Without Disease Progression During 1L Treatment With Aromatase Inhibitor+ CDK4/6 Inhibitor- A ctDNA Guided Early Switch Study
Brief Title: Phase III Study to Assess AZD9833+ CDK4/6 Inhibitor in HR+/HER2-MBC With Detectable ESR1m Before Progression (SERENA-6)
Acronym: SERENA-6
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: D8534C00001; 2023-503990-39-00 (Other: EU CT number); 2021-000546-17 (EudraCT Number)
Record Dates: First submitted 2021-06-30; First posted 2021-07-16 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2025-12

CONDITIONS: ER-Positive HER2-Negative Breast Cancer
Keywords: Metastatic; Breast Neoplasms; Neoplasms by Site; Neoplasms; Breast Diseases; Physiological Effects of Drugs; Randomised; Multicentre; Double-Blind; Phase III; AZD9833; Next Generation Oral SERD; Anastrozole; Letrozole; Palbociclib; Abemaciclib; Ribociclib; Antagonists; Antineoplastic Agents; Estrogen Receptor Antagonists; Hormone Antagonists; camizestrant; ESR1m; Switch Treatment; Endocrine Therapy; Endocrine Resistance
MeSH Terms: conditions — Neoplasm Metastasis; Breast Neoplasms; Neoplasms by Site; Neoplasms; Breast Diseases | interventions — AZD9833; Anastrozole; Letrozole; palbociclib; abemaciclib; Gonadotropin-Releasing Hormone; ribociclib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- AZD9833 + palbociclib, abemaciclib or ribociclib (Experimental): The patients will receive AZD9833 (75 mg, PO, once daily) + palbociclib (PO, once daily, 125, 100 or 75 mg for 21 consecutive days followed by 7 days off treatment), abemaciclib (PO, twice daily, 150,100 or 50 mg) or ribociclib (To Be Determined, PO, once daily for 21 consecutive days followed by 7 days off treatment) + anastrozole placebo (PO, once daily) or letrozole placebo (PO, once daily)
  Interventions: Drug: AZD9833; Drug: Anastrozole placebo; Drug: Letrozole placebo; Drug: Palbociclib; Drug: Abemaciclib; Drug: Luteinizing hormone-releasing hormone (LHRH) agonist; Drug: Ribociclib
- Anastrozole or letrozole + palbociclib, abemaciclib or ribociclib (Active Comparator): The patients will recieve anastrozole (1 mg, PO, once daily) or letrozole (2.5 mg, PO, once daily) + palbociclib (PO, once daily, 125, 100 or 75 mg for 21 consecutive days followed by 7 days off treatment), abemaciclib (PO, twice daily, 150, 100 or 50 mg) or ribociclib (To Be Determined, PO, once daily for 21 consecutive days followed by 7 days off treatment) + AZD9833 placebo (PO, once daily)
  Interventions: Drug: AZD9833 Placebo; Drug: Anastrozole; Drug: Letrozole; Drug: Palbociclib; Drug: Abemaciclib; Drug: Luteinizing hormone-releasing hormone (LHRH) agonist; Drug: Ribociclib

INTERVENTIONS:
Drug: AZD9833 — Dosage formulation: AZD9833 tablets will be administered orally
  Arms: AZD9833 + palbociclib, abemaciclib or ribociclib
Drug: AZD9833 Placebo — Dosage formulation: AZD9833 placebo tablets will be administrated orally.
  Arms: Anastrozole or letrozole + palbociclib, abemaciclib or ribociclib
Drug: Anastrozole — Dosage formulation: anastrozole tablets will be administered orally.
  Arms: Anastrozole or letrozole + palbociclib, abemaciclib or ribociclib
Drug: Anastrozole placebo — Dosage formulation: anastrozole placebo tablets will be administrated orally.
  Arms: AZD9833 + palbociclib, abemaciclib or ribociclib
Drug: Letrozole — Dosage formulation: letrozole tablets will be administered orally.
  Arms: Anastrozole or letrozole + palbociclib, abemaciclib or ribociclib
Drug: Letrozole placebo — Dosage formulation: letrozole placebo tablets will be administered orally.
  Arms: AZD9833 + palbociclib, abemaciclib or ribociclib
Drug: Palbociclib — Dosage formulation: palbociclib tablets/capsules will be administered orally
Drug: Abemaciclib — Dosage formulation: abemaciclib tablets will be administered orally
Drug: Luteinizing hormone-releasing hormone (LHRH) agonist — Men (when medically applicable) and pre- or peri-menopausal women are required to receive a monthly LHRH agonist.
Drug: Ribociclib — Dosage formulation: ribociclib tablets will be administered orally

SUMMARY:
The study is intended to show superiority of AZD9833 in combination with CDK4/6 inhibitor (palbociclib, abemaciclib or ribociclib) versus aromatase inhibitors (anastrozole or letrozole) in combination with CDK4/6 inhibitor in patients with hormone receptor-positive (HR-positive), human epidermal growth factor receptor 2-negative (HER2-negative) metastatic breast cancer with detectable ESR1 mutation.

DETAILED DESCRIPTION:
Breast cancer is the most common type of cancer among women. In people with breast cancer, the body is not able to control the growth of some cells. These extra cells can form tumors in the breast. When tumor cells move to different parts of the body this is called advanced cancer. Researchers are looking for better ways to treat advanced breast cancer.

This trial will look at six drugs: palbociclib, abemaciclib, ribociclib, letrozole, anastrozole, and AZD9833. AZD9833 is the trial drug, and is the only drug not yet approved for use. Palbociclib, abemaciclib and ribociclib work in the same way and are a type of cancer drug called a CDK4/6 inhibitor. Letrozole and anastrozole work in the same way and are both a type of cancer drug called an aromatase inhibitor (AI). CDK4/6 inhibitors and AIs work together to block the tumor's ability to grow. These drugs have been approved for combined use in people with advanced breast cancer that is HR-positive and HER2-negative. But if people get mutations in the ESR1 gene, it can make the AI and CDK4/6 inhibitor treatment work less well.

The trial drug, AZD9833, is designed to work with a CDK4/6 inhibitor in the same way that an AI does. Researchers think that AZD9833 might work better with a CDK4/6 inhibitor than an AI does in people who get mutations in their ESR1 gene.

Participants in this trial will have already been receiving one of the following combinations of a CDK4/6 inhibitor and an AI:

* palbociclib + anastrozole
* palbociclib + letrozole
* abemaciclib + anastrozole
* abemaciclib + letrozole
* ribociclib + anastrozole
* ribociclib + letrozole

During the trial, participants will remain on the same CDK4/6 inhibitor that they were taking before the trial.

In this trial, the researchers want to find out how well switching a participant with an ESR1 gene mutation from an AI (letrozole or anastrozole) to AZD9833 works in the treatment of advanced breast cancer that is HR-positive and HER2-negative.

The researchers will look at which trial treatment helps the participants live longer with the cancer before it gets worse.

The researchers also want to know more about how safe AZD9833 is.

The trial participants will be split into 2 groups:

* Participants in Group A will receive AZD9833, a CDK4/6 inhibitor, and a placebo
* Participants in Group B will receive an AI, a CDK4/6 inhibitor, and a placebo

A placebo looks like a treatment but does not have any medicine in it.

A computer program will be used to randomly choose the treatments each participant gets. This helps make sure the groups are chosen fairly. Researchers do this so that comparing the results of each treatment will be as accurate as possible.

The participants will take their trial treatments over 28-day cycles, with a placebo and either AZD9833 or an AI taken once daily by mouth for all 28 days. If the participant is taking abemaciclib, they will take it twice daily by mouth for all 28 days. If the participant is taking palbociclib or ribociclib, they will take it once daily by mouth for 21 days and then stop taking it for the final 7 days of the cycle. The participant will then repeat the 28-day cycle receiving the trial treatment in the same way for as long as they are in the trial.

Participants will visit their trial site regularly throughout the trial. At these visits, the trial doctors will check the health of the participants. They will also take blood samples and do scans of the participants' tumors.

Participants will take their trial treatment until their cancer gets worse or they decide to leave the trial.

ELIGIBILITY:
INCLUSION CRITERIA:

INFORMATION FOR TRIAL PARTICIPANTS - Participants can join the trial if they:

* Have advanced breast cancer that is not able to be treated with surgery or radiation;
* Have an ESR1 mutation in their cancer;
* Have breast cancer that is HR-positive and HER2-negative;
* Are currently being treated with a CDK4/6 inhibitor and an AI and have been taking these drugs for at least 6 months;
* Have not had their cancer get worse after taking an AI and CDK4/6 inhibitor;
* Are able to do their daily activities;
* Are at least 18.

Full list of inclusion criteria:

* Proven diagnosis of adenocarcinoma of the breast with evidence of locoregionally recurrent or metastatic disease not amenable to resection or radiation therapy with curative intent;
* Documentation of histologically confirmed diagnosis of estrogen receptor positive (ER+) /HER2- breast cancer based on local laboratory results;
* Currently on AI (letrozole or anastrozole) + CDK4/6 inhibitor (palbociclib, abemaciclib or ribociclib) ± LHRH as the initial endocrine based treatment for advanced disease;
* Eastern Cooperative Oncology Group performance status of 0 or 1;
* ESR1m detected by central testing of ctDNA with Guardant360® CDx;
* Willingness and ability to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures;
* Adequate organ and marrow function.

EXCLUSION CRITERIA:

INFORMATION FOR TRIAL PARTICIPANTS - Participants cannot join the trial if they:

* Had certain types of tumors in the past that may come back;
* Are currently taking any other treatments for their cancer or other conditions including hormone replacements, medications, or supplements that could interfere with the trial treatment;
* Have or have had any major health problem, infection, or recent surgery that could make it difficult or dangerous to participate in this trial.

Full list of exclusion criteria:

* Advanced, symptomatic, visceral spread, that are at risk of life-threatening complications in the short term;
* Known active uncontrolled or symptomatic CNS metastases, carcinomatous meningitis, or leptomeningeal disease;
* Any evidence of severe or uncontrolled systemic diseases which, in the investigator's opinion, makes it undesirable for the participant to participate in the study or that would jeopardize compliance with the protocol;
* Patient with known or family history of severe heart disease;
* Previous treatment with AZD9833, investigational SERDs or fulvestrant;
* Currently pregnant (confirmed with positive pregnancy test) or breastfeeding;
* Persistent non-haematological toxicities (CTCAE Grade > 2) caused by CDK4/6 inhibitor and/or AI treatment.

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 315 (Actual)
Dates: Start 2021-06-30 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2027-11-26 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) assessed by the Investigator as defined by response evaluation criteria in solid tumors (RECIST version 1.1) | From randomization until the earlier of the progression event or death (approximately 2 years)
  PFS is defined as the time from randomization to objective disease progression (as assessed by RECIST 1.1) or death.

SECONDARY OUTCOMES:
Progression-free survival 2 (PFS2) | From randomization to the earliest of the progression event (following the initial progression), subsequent to first subsequent therapy or death (approximately 3.5 years)
  PFS2 is defined as the time from the randomisation to the earliest of the progression event (following the initial progression), subsequent to first subsequent therapy or death.
Overall survival (OS) | From randomization until the date of death due to any cause (approximately 5 years)
  The OS is defined as the time from randomization to death due to any cause.
Chemotherapy free survival | From randomization until the earlier of the start date of chemotherapy or death due to any cause (approximately 5 years)
  Time to chemotherapy is defined as the time from randomization until the earlier of the start date of chemotherapy or death due to any cause.
Objective response rate (ORR) assessed by the Investigator as defined by RECIST version 1.1 | From randomization until a response or in the absence of a response from randomization up until progression, or the last evaluable assessment in the absence of progression (approximately 5 years)
  ORR is defined as the proportion of patients who have a complete response (CR) or partial response (PR), as determined by the investigator at local site per RECIST 1.1.
Clinical benefit rate at 24 weeks (CBR24) | At least 23 weeks after randomisation for each patient (1 week window for RECIST assessment)
  CBR at 24 weeks is defined as the percentage of participants who have a complete response (CR) or partial response or who have stable disease (SD) per RECIST 1.1 as assessed by the investigator at local site for At least 23 weeks after randomisation for each patient to allow for an early assessment within the assessment window (1 week window for RECIST assessment)
Change from baseline in EORTC QLQ-C30 scale scores | From baseline until second progression (approximately 5 years)
  Change from baseline in scales scores of the European Organisation for the Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-C30). Scale scores range from 0-100. For functioning and global health status/ QoL scales, higher scores indicate better functioning or global health status/QoL. For symptom scales, higher scores indicate greater symptom burden.
Change from baseline in EORTC QLQ-BR23 scale scores | From baseline until second progression (approximately 5 years)
  Change from baseline in scales scores of the European Organisation for the Research and Treatment of Cancer Quality of Life Questionnaire Breast Cancer Module (EORTC QLQ-BR23). Scale scores range from 0-100. For functioning scales, higher scores indicate better functioning. For symptom scales, higher scores indicate greater symptom burden.
Plasma concentration of AZD9833 at specified timepoints | on Day 15 for each patient
  To assess the steady state PK of AZD9833 in combination with palbociclib or abemaciclib in all participants who receive at least one dose of AZD9833 per the protocol, for whom there are at least one reportable PK concentration.

CONTACTS AND LOCATIONS:
Locations (223):
- United States (60):
  - Research Site, Phoenix, Arizona
  - Research Site, Hot Springs, Arkansas
  - Research Site, Little Rock, Arkansas
  - Research Site, Long Beach, California
  - Research Site, San Diego, California
  - Research Site, Santa Rosa, California
  - Research Site, Grand Junction, Colorado
  - Research Site, Lone Tree, Colorado
  - Research Site, Fort Myers, Florida
  - Research Site, Jacksonville, Florida
  - Research Site, St. Petersburg, Florida
  - Research Site, Atlanta, Georgia
  - Research Site, Park Ridge, Illinois
  - Research Site, Fort Wayne, Indiana
  - Research Site, Indianapolis, Indiana
  - Research Site, Baltimore, Maryland
  - Research Site, Boston, Massachusetts
  - Research Site, Fairhaven, Massachusetts
  - Research Site, Foxborough, Massachusetts
  - Research Site, Milford, Massachusetts
  - Research Site, South Weymouth, Massachusetts
  - Research Site, Detroit, Michigan
  - Research Site, Grand Rapids, Michigan
  - Research Site, Rochester, Minnesota
  - Research Site, Oxford, Mississippi
  - Research Site, Kansas City, Missouri
  - Research Site, St Louis, Missouri
  - Research Site, Billings, Montana
  - Research Site, Omaha, Nebraska
  - Research Site, Camden, New Jersey
  - Research Site, Ridgewood, New Jersey
  - Research Site, Brooklyn, New York
  - Research Site, East Syracuse, New York
  - Research Site, New Hyde Park, New York
  - Research Site, New York, New York
  - Research Site, Shirley, New York
  - Research Site, Goldsboro, North Carolina
  - Research Site, Canton, Ohio
  - Research Site, Cincinnati, Ohio
  - Research Site, Columbus, Ohio
  - Research Site, Portland, Oregon
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Pittsburgh, Pennsylvania
  - Research Site, York, Pennsylvania
  - Research Site, Greenville, South Carolina
  - Research Site, West Columbia, South Carolina
  - Research Site, Knoxville, Tennessee
  - Research Site, Memphis, Tennessee
  - Research Site, Nashville, Tennessee
  - Research Site, Bedford, Texas
  - Research Site, Dallas, Texas
  - Research Site, Houston, Texas
  - Research Site, Irving, Texas
  - Research Site, Longview, Texas
  - Research Site, San Antonio, Texas
  - Research Site, Salt Lake City, Utah
  - Research Site, Midlothian, Virginia
  - Research Site, Norfolk, Virginia
  - Research Site, Tacoma, Washington
  - Research Site, Waukesha, Wisconsin
- Australia (2):
  - Research Site, Birtinya
  - Research Site, Darlinghurst
- Austria (4):
  - Research Site, Graz
  - Research Site, Innsbruck
  - Research Site, Salzburg
  - Research Site, Vienna
- Belgium (3):
  - Research Site, Leuven
  - Research Site, Liège
  - Research Site, Namur
- Bulgaria (5):
  - Research Site, Haskovo
  - Research Site, Panagyurishte
  - Research Site, Pleven
  - Research Site, Plovdiv
  - Research Site, Sofia
- Canada (6):
  - Research Site, Calgary, Alberta
  - Research Site, Vancouver, British Columbia
  - Research Site, Ottawa, Ontario
  - Research Site, Lévis, Quebec
  - Research Site, Montreal, Quebec
  - Research Site, Québec, Quebec
- France (19):
  - Research Site, Avignon
  - Research Site, Brest
  - Research Site, Clermont-Ferrand
  - Research Site, Dijon
  - Research Site, Limoges
  - Research Site, Lorient
  - Research Site, Lyon
  - Research Site, Marseille
  - Research Site, Metz-Tessy
  - Research Site, Nîmes
  - Research Site, Paris
  - Research Site, Rouen
  - Research Site, Saint-Cloud
  - Research Site, Saint-Herblain
  - Research Site, Toulouse
  - Research Site, Tours
  - Research Site, Vandœuvre-lès-Nancy
  - Research Site, Vantoux
  - Research Site, Villejuif
- Germany (21):
  - Research Site, Ansbach
  - Research Site, Aschaffenburg
  - Research Site, Augsburg
  - Research Site, Bonn
  - Research Site, Chemnitz
  - Research Site, Dresden
  - Research Site, Erlangen
  - Research Site, Essen
  - Research Site, Freiburg im Breisgau
  - Research Site, Immenstadt im Allgäu
  - Research Site, Koblenz
  - Research Site, Leipzig
  - Research Site, Mannheim
  - Research Site, München
  - Research Site, Paderborn
  - Research Site, Ratingen
  - Research Site, Ravensburg
  - Research Site, Regensburg
  - Research Site, Stade
  - Research Site, Tübingen
  - Research Site, Ulm
- Hungary (5):
  - Research Site, Budapest
  - Research Site, Miskolc
  - Research Site, Szekszárd
  - Research Site, Szolnok
  - Research Site, Zalaegerszeg
- Israel (5):
  - Research Site, Beersheba
  - Research Site, Haifa
  - Research Site, Jerusalem
  - Research Site, Petah Tikva
  - Research Site, Ramat Gan
- Italy (10):
  - Research Site, Bergamo
  - Research Site, Bologna
  - Research Site, Florence
  - Research Site, Meldola
  - Research Site, Milan
  - Research Site, Misterbianco
  - Research Site, Napoli
  - Research Site, Padua
  - Research Site, Roma
  - Research Site, Rozzano
- Japan (19):
  - Research Site, Chiba
  - Research Site, Chūōku
  - Research Site, Hidaka-shi
  - Research Site, Hirakata-shi
  - Research Site, Kitaadachi-gun
  - Research Site, Kōtoku
  - Research Site, Kumamoto
  - Research Site, Matsuyama
  - Research Site, Nagoya
  - Research Site, Niigata
  - Research Site, Osaka
  - Research Site, Ota-shi
  - Research Site, Sapporo
  - Research Site, Shinagawa-ku
  - Research Site, Shinjuku-ku
  - Research Site, Takasaki-shi
  - Research Site, Takatsuki-shi
  - Research Site, Tsukuba
  - Research Site, Yokohama
- Norway (2):
  - Research Site, Drammen
  - Research Site, Oslo
- Poland (8):
  - Research Site, Bydgoszcz
  - Research Site, Gdynia
  - Research Site, Koszalin
  - Research Site, Lodz
  - Research Site, Poznan
  - Research Site, Rzeszów
  - Research Site, Tomaszów Mazowiecki
  - Research Site, Warsaw
- Portugal (5):
  - Research Site, Guimarães
  - Research Site, Lisbon
  - Research Site, Loures
  - Research Site, Porto
  - Research Site, Vila Nova de Gaia
- Russia (4):
  - Research Site, Moscow
  - Research Site, Nizhny Novgorod
  - Research Site, Podolsk
  - Research Site, Saint Petersburg
- Slovakia (5):
  - Research Site, Banská Bystrica
  - Research Site, Bratislava
  - Research Site, Košice
  - Research Site, Michalovce
  - Research Site, Partizánske
- South Korea (5):
  - Research Site, Cheonan-si
  - Research Site, Daegu
  - Research Site, Goyang-si
  - Research Site, Seongnam-si
  - Research Site, Seoul
- Spain (10):
  - Research Site, A Coruña
  - Research Site, Badalona
  - Research Site, Barcelona
  - Research Site, L'Hospitalet de Llobregat
  - Research Site, Madrid
  - Research Site, Málaga
  - Research Site, Murcia
  - Research Site, Sant Joan Despí
  - Research Site, Seville
  - Research Site, Valencia
- Switzerland (3):
  - Research Site, Bern
  - Research Site, Chur
  - Research Site, Winterthur
- Taiwan (5):
  - Research Site, Kaohsiung City
  - Research Site, Taichung
  - Research Site, Tainan
  - Research Site, Taipei
  - Research Site, Taoyuan District
- Turkey (Türkiye) (6):
  - Research Site, Adana
  - Research Site, Ankara
  - Research Site, Izmir
  - Research Site, Kadıkoy/Istanbul
  - Research Site, Karşıyaka
  - Research Site, Kayseri
- United Kingdom (11):
  - Research Site, Blackpool
  - Research Site, Cambridge
  - Research Site, London
  - Research Site, Manchester
  - Research Site, Newport
  - Research Site, Nottingham
  - Research Site, Portsmouth
  - Research Site, Reading
  - Research Site, Sheffield
  - Research Site, Sutton
  - Research Site, Taunton

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the deidentified individual patient-level data in an approved sponsored tool. Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- [Derived] Bidard FC, Mayer EL, Park YH, Janni W, Ma C, Cristofanilli M, Bianchini G, Kalinsky K, Iwata H, Chia S, Fasching PA, Brufsky A, Nowecki Z, Pascual J, Moreau L, Chen SC, Karadurmus N, Gal-Yam EN, Jung KH, Pernas S, McClain S, He W, Klinowska T, Huang-Bartlett C, Turner NC; SERENA-6 Study Group. First-Line Camizestrant for Emerging ESR1-Mutated Advanced Breast Cancer. N Engl J Med. 2025 Aug 7;393(6):569-580. doi: 10.1056/NEJMoa2502929. Epub 2025 Jun 1. PMID 40454637
- [Derived] Turner N, Huang-Bartlett C, Kalinsky K, Cristofanilli M, Bianchini G, Chia S, Iwata H, Janni W, Ma CX, Mayer EL, Park YH, Fox S, Liu X, McClain S, Bidard FC. Design of SERENA-6, a phase III switching trial of camizestrant in ESR1-mutant breast cancer during first-line treatment. Future Oncol. 2023 Mar;19(8):559-573. doi: 10.2217/fon-2022-1196. Epub 2023 Apr 18. PMID 37070653
- See also: Breast Cancer Study Locator details (for US) — https://www.breastcancerstudylocator.com/trial/listing/296201